CLINICAL TRIAL: NCT01140828
Title: A Double-blind Randomized Placebo Controlled Trial of Rabeprazole for Prevention of NSAID-associated Dyspepsia and Gastroduodenal Injury
Brief Title: A Study of Rabeprazole for Prevention of Non Steroidal Anti-inflammatory Drug -Associated Gastroduodenal Injury
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Francis KL Chan, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RAN Study
Record Dates: First submitted 2010-06-09; First posted 2010-06-10 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Osteoarthritis; Arthritis, Rheumatoid; Dyspepsia
Keywords: Arthritis; Bone pain; dyspepsia
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Dyspepsia; Arthritis | interventions — Rabeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rabeprazole (Active Comparator): Rabeprazole
  Interventions: Drug: Rabeprazole
- Rabeprazole Placebo (Placebo Comparator): Rabeprazole Placebo
  Interventions: Drug: Rabeprazole Placebo

INTERVENTIONS:
Drug: Rabeprazole — Rabeprazole 20mg once daily
  Other Names: Pariet
  Arms: Rabeprazole
Drug: Rabeprazole Placebo — one tab once daily
  Other Names: Pariet Placebo
  Arms: Rabeprazole Placebo

SUMMARY:
The aim of this study is to determine whether rabeprazole is superior to placebo in preventing dyspepsia and gastroduodenal injury in subjects with osteoarthritis (OA) and/or rheumatoid arthritis (RA) and/or bone pain.

DETAILED DESCRIPTION:
Non steroidal anti-inflammatory drugs (NSAIDs) are well known to increase the risk of gastroduodenal (GD) ulcer and its complications. Up to 40% of average-risk NSAID users suffer from dyspepsia without endoscopic evidence of gastroduodenal injury. It results a significant loss of productivity and impairment of Quality of Life (QoL). Proton pump inhibitors (PPIs) have been shown to be effective in preventing and reducing NSAID-induced GD injury. PPIs are believed to have a class effect but Rabeprazole, the least expensive PPI, is grossly under-utilized in this area .

Current Hospital Authority (HA) guidelines, however, only endorse the use of PPI in patients at high risk of ulcer bleeding. Since NSAID-induced dyspepsia is not an indication for PPI according to HA guidelines, those patients do not receive PPI for treatment.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient or inpatient subjects with a clinical diagnosis of OA or RA or any bone pain
* Subjects expected to require regular anti-inflammatory therapy for arthritis symptom management
* Subjects should have no history of peptic ulcer complications
* Screening tests are negative for H pylori
* Subjects who test positive can be re-screened after eradication of H. pylori

Exclusion Criteria:

* History of gastrointestinal (GI) hemorrhage
* History of gastric or duodenal surgery
* Presence of erosive esophagitis, gastric-outlet obstruction
* Likelihood of requiring treatment during the study with drugs not permitted by the protocol
* Impaired hepatic function (SGPT (ALT) or serum glutamate oxaloacetate transaminase (SGOT) (AST) > 2 x upper limit of normal) or renal function (serum creatinine > 200 umol/l)
* Any other condition or baseline finding which, in the investigator's judgment, might increase risk to the subject or decrease the chance of obtaining satisfactory data to achieve study objectives
* Anemia with Hb < 10 g/dL
* Suspected or clinical diagnosis of inflammatory bowel disease
* Congestive heart failure (NYHA class III- IV)
* Subjects considered to have a requirement for continued use of:

  * Corticosteroids (dose equivalent of prednisolone/ prednisone >10mg daily stable dose)
  * disease-modifying antirheumatic drug (DMARDs) (unless stable dose for ≥ 12 weeks)
  * Iron replacement therapy (a dose > 15mg elemental iron/day)
  * Iron replacement therapy (a dose > 15mg elemental iron/day) or supplements for deficiency prevention (a dose ≤ 15mg elemental iron/day) due to anemia or any other reason
  * Double anti-platelet therapy (e.g. aspirin + Plavix)
  * Anti-coagulants
  * Anti-ulcer medications, e.g. sucralfate, H2 receptor antagonists (H2RAs), misoprostol, PPIs other than study medications
  * Sucralfate, misoprostol or regular H2 receptor antagonists (H2RAs) (> 3 days/week)
  * COX-2 inhibitors
  * anti-ulcer medications or COX-2 selective inhibitor at screening allowed if treatments discontinued at this time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2009-05; Primary Completion 2012-10 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
12-week cumulative incidence of gastric/duodenal ulcer, >10 erosions or severe dyspepsia | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Francis K Chan, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong, China